CLINICAL TRIAL: NCT00900562
Title: Phase II Clinical and Pharmacokinetic Trial of PM00104 (Zalypsis®) in Patients With Advanced and/or Metastatic Endometrial or Cervical Cancer Previously Treated With One Line of Systemic Chemotherapy
Brief Title: Clinical Trial of PM00104 (Zalypsis®) in Patients With Advanced and/or Metastatic Endometrial or Cervical Cancer Previously Treated With One Line of Systemic Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow and poor recruitment.
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM104-B-001-09
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Results first posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-07

CONDITIONS: Uterine Cervical Cancer; Endometrial Cancer
Keywords: Zalypsis; Cancer; Endometrial; Uterine Cervical; PharmaMar
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Neoplasms | interventions — PM 00104

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Zalypsis (PM00104)
  Interventions: Drug: Zalypsis ( PM00104)

INTERVENTIONS:
Drug: Zalypsis ( PM00104) — Zalypsis (PM00104) (2.5 mg/vial) is provided as a powder for concentrate for solution for infusion

SUMMARY:
This study is a phase II clinical and pharmacokinetic trial of PM00104 (Zalypsis®) in patients with advanced and/or metastatic endometrial or cervical cancer previously treated with one line of systemic chemotherapy to evaluate the antitumor activity and to determine the safety profile, the pharmacokinetic profile and the pharmacogenomic profile.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent, obtained from the patient before the beginning of any specific study procedures.
2. Group 1 (endometrial cancer):

   * Histologically confirmed advanced and/or metastatic endometrial cancer (any grade, including endometrioid, clear cell, serous and mixed types) with documented disease progression as per RECIST at study entry.
   * Patients must have failed one prior systemic chemotherapy line for advanced/metastatic disease (excluding chemosensitizing chemotherapy); prior hormone therapy and biological therapy are allowed.
3. Group 2 (cervical cancer):

   * Histologically confirmed advanced and/or metastatic cervical cancer with documented disease progression as per RECIST at study entry.
   * Patients must have failed one prior systemic chemotherapy line for advanced/metastatic disease (excluding chemosensitizing chemotherapy); prior hormone therapy and biological therapy are allowed.
4. Complete recovery from the effects of prior radiotherapy and from any drug-related adverse events (AEs) derived from previous treatments, excluding alopecia and grade 1 peripheral neuropathy according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCICTCAE, v.3.0).
5. At least one measurable lesion ("target lesion" according to the RECIST), located in a non-irradiated area and adequately measured less than four weeks before study entry. Tumors within a previously irradiated field will be designated as "nontarget" lesions unless progression is clearly documented or biopsy proven.
6. Age ≥ 18 years.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 1.
8. Life expectancy ≥ 3 months.
9. Appropriate bone marrow reserve, renal and hepatic functions:

   * Platelet count ≥ 100 x 109/l, hemoglobin ≥ 9 g/dl and absolute neutrophil count (ANC) ≥ 1.5 x 109/l.
   * Alkaline phosphatase (AP) ≤ 2.5 x upper limit of normality (ULN) (≤ 5 x ULN in case of extensive bone metastases).
   * Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN in case of hepatic metastases).
   * Total bilirubin ≤ 1.5 x ULN, unless due to Gilbert's syndrome.
   * Renal function: patients with calculated creatinine clearance (using Cockcroft and Gault formula) ≥ 30 ml/min.
   * Albumin ≥ 2.5 g/dl.
10. Left ventricular ejection fraction (LVEF) within normal limits (LVEF of at least 50%).
11. Women of childbearing potential must have a negative serum pregnancy test before study entry. In case of childbearing potential, the patients and their partners must agree to use a medically acceptable method of contraception.

Exclusion Criteria:

1. Prior therapy with PM00104.
2. Uterine sarcomas, adenosarcoma, and malignant Mullerian tumors.
3. Cervical neuroendocrine or small cell carcinomas, nonepithelial cervical neoplasms such as sarcomas.
4. Patients who have isolated recurrences (vaginal, pelvic or paraaortic) potentially curative with radiation therapy or surgery.
5. Pregnant or lactating women, or in case of childbearing potential, women not using an appropriate contraceptive method.
6. Less than three weeks from prior radiation therapy, biological therapy or chemotherapy, AND

   * Less than six weeks from prior nitrosourea, mitomycin C, high-dose chemotherapy or radiotherapy involving the whole pelvis or over 50% of the spine, provided that acute effects of radiation treatment have resolved.
   * Hormonal therapy and palliative radiation therapy (i.e., for control of pain from bone metastases) must be discontinued before study entry.
7. Group 1 (endometrial cancer): more than one line of prior systemic chemotherapy for advanced/metastatic disease (excluding chemosensitizing chemotherapy), but not less than three weeks before.
8. Group 2 (cervical cancer): more than one line of prior systemic chemotherapy for advanced/metastatic disease (excluding chemosensitizing chemotherapy, but not less than three weeks before.
9. Patients with a prior invasive malignancy (except nonmelanoma skin cancer) who have had any evidence of disease within the last five years or whose prior malignancy treatment contraindicates the current protocol therapy.
10. Patients with serious non-healing wound, ulcer, or bone fracture.

    * This includes history of: abdominal fistula, gastrointestinal perforation or intra-abdominal abscess for which an interval of three to six months must pass before study entry.
    * In addition, the patient must have undergone correction (or spontaneous healing) of the perforation/fistula and/or the underlying process causing the fistula/perforation.
    * Patients with granulating incisions healing by secondary intention with no evidence of fascial dehiscence or infection are eligible but require weekly wound examinations.
11. Evidence of progressive or symptomatic central nervous system (CNS) metastases or leptomeningeal metastases.
12. Other diseases or serious conditions:

    * Increased cardiac risk as defined by:

      * Unstable angina or myocardial infarction within 12 months before inclusion in the study.
      * New York Heart Association (NYHA) grade II or greater congestive heart failure.
      * Symptomatic arrhythmia or any arrhythmia requiring ongoing treatment.
      * Abnormal electrocardiogram (ECG), i.e., patients with the following are excluded: QT prolongation - QTc > 480 msec; signs of cardiac enlargement or hypertrophy; bundle branch block; partial blocks;signs of ischemia or necrosis, and Wolff Parkinson White patterns.
      * History or presence of valvular heart disease.
      * Uncontrolled arterial hypertension despite optimal medical therapy.
      * Previous mediastinal radiotherapy.
      * Previous treatment with doxorubicin at cumulative doses exceeding 400 mg/m2.
    * History of significant neurological or psychiatric disorders.
    * Active infection requiring systemic treatment.
    * Significant non-neoplastic liver disease (e.g., cirrhosis, active chronic hepatitis).
    * Immunocompromised patients, including those known to be infected with the human immunodeficiency virus (HIV).
    * Uncontrolled (i.e., requiring relevant changes in medication within the last month or hospital admission within the last three months) endocrine diseases (e.g., diabetes mellitus, hypo- or hyperthyroidism, adrenal disorder).
13. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in the study. The investigator should feel free to consult the Study Coordinator or the Sponsor for uncertainty in this regard.
14. Limitation of the patient's ability to comply with the treatment or to follow-up at a participating center. Patients enrolled into this trial must be treated and followed at a participating center.
15. Treatment with any investigational product within 30 days prior to inclusion in the study.
16. Known hypersensitivity to any component of PM00104.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - UNM (University of New Mexico) Cancer Center, Albuquerque, New Mexico
  - OU Cancer Institute, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Endometrial Cancer: 12 patients were recruited and treated at 4 sites in the US. Patients participated between 14/08/2009 (first consent signed (CS)) and 22/2/2010 (last CS). The first dose was administered on 26/08/2009 and the last dose on 2/4/2010.
  Cervical Cancer: 7 patients were recruited and treated at 3 sites in the US. Patients participated in the study between 19/8/2009 (first CS) and 22/12/2010 (last CS). The first dose was administered on 26/10/2009 and the last dose on 10/03/2011
Groups:
- Endometrial Cancer: Patients with Endometrial Cancer. A treatment cycle consisted of the administration of i.v. 1-hour infusions of PM00104 on Day 1, Day 8 and Day 15, and all study evaluations done before the next cycle. Treatment cycles were to be repeated every four weeks.
  Study treatment was administered to patients by a central catheter and by specialized on-site study personnel. A central catheter was mandatory as some cases of infusion site reactions were observed in the phase I trials
- Cervical Cancer: Patients with Cervical Cancer A treatment cycle consisted of the administration of i.v. 1-hour infusions of PM00104 on Day 1, Day 8 and Day 15, and all study evaluations done before the next cycle. Treatment cycles were to be repeated every four weeks.
  Study treatment was administered to patients by a central catheter and by specialized on-site study personnel. A central catheter was mandatory as some cases of infusion site reactions were observed in the phase I trials
Period: Overall Study
Arm/Group | Endometrial Cancer | Cervical Cancer
Started | 12 | 7
Completed | 0 | 0
Not Completed | 12 | 7
Not completed — Progressive disease | 9 | 5
Not completed — Toxicity | 1 | 0
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Unrelated adverse event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endometrial Cancer | Cervical Cancer | Total
Number analyzed (Participants) | 12 | 7 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 16
  >=65 years | 3 | 0 | 3
Age, Continuous [Median (Full Range); unit: years] | 61.5 [51 to 69] | 38 [29 to 62] | 59 [29 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 4 | 10
  Hispanic | 3 | 0 | 3
  African American | 0 | 1 | 1
  Black | 3 | 1 | 4
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 7 | 19
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status, ECOG PS 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. Dead
  Participants
    0 | 5 | 1 | 6
    1 | 7 | 6 | 13
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 0 | 1 | 1
  Adenosquamous | 0 | 3 | 3
  Clear cell | 1 | 0 | 1
  Endometrioid | 4 | 0 | 4
  Mixed | 3 | 0 | 3
  Other | 1 | 1 | 2
  Papillary serous | 3 | 0 | 3
  Squamous cell carcinoma | 0 | 2 | 2
Extent of disease [Count of Participants; unit: Participants]
  Metastatic | 10 | 7 | 17
  Locally advanced | 2 | 0 | 2
Histology grade [Count of Participants; unit: Participants] — Low grade or grade I tumors are well-differentiated. This means that the tumor cells are organized and look more like normal tissue.
  High grade or grade III tumor cells are poorly differentiated. This means that the tumor cells don't look like normal cells. They're disorganized under the microscope and tend to grow and spread faster than grade I tumors.
  Cancer cells that don't look well-differentiated or poorly differentiated are called moderately differentiated, or grade II.
  Participants
    Poorly differentiated | 10 | 6 | 16
    Moderately differentiated | 1 | 1 | 2
    Unknown | 1 | 0 | 1
Sites involved [Count of Participants; unit: Participants]
  1 | 6 | 1 | 7
  2 | 2 | 2 | 4
  3 | 2 | 2 | 4
  >3 | 2 | 2 | 4
Time from diagnosis to first infusion [Median (Full Range); unit: months] | 18.2 [7.5 to 48.8] | 10.7 [6.9 to 91.3] | 16.6 [6.9 to 91.3]
Time from last progression to first infusion [Median (Full Range); unit: months] | 0.9 [0.1 to 5.5] | 0.8 [0.4 to 6.4] | 0.8 [0.1 to 6.4]
Prior Surgery [Count of Participants; unit: Participants] | 11 | 6 | 17
Prior Systemic anticancer therapy [Count of Participants; unit: Participants] | 12 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate defined as the percentage of patients with either complete response (CR) or partial response (PR) according to RECIST v.1.0.
  CR, complete response: disappearance of all lesions; PD, disease progression: ≥10% increase in target lesion size and does not meet tumor density criteria of PR density; PR, partial response: ≥10% decrease in target lesion size or ≥15% decrease in tumor density; SD, stable disease: none of the CR, PR, or PD criteria met; RECIST, Response Evaluation Criteria in Solid Tumors
Time Frame: At baseline and every other cycle (± 1 week) until evidence of PD, up to 2 years
Population: Two patients were not evaluable for efficacy: One patient received only one PM00104 infusion in Cycle 1 and had to be withdrawn from the study due to a troponin I increase, which occurred seven days after the first infusion of PM00104 and was considered serious (SAE) and related to PM00104; One patient only received one PM00104 infusion and was withdrawn from the study due to drug-unrelated marantic endocarditis
Measure: Count of Participants; unit: Participants
Arm/Group | Endometrial Cancer | Cervical Cancer
Number analyzed (Participants) | 10 | 7
Participants | 0 | 0

2. Secondary Outcome: Best Tumor Response
Description: Best tumor response was defined as the best response achieved during the study according to RECIST v1.0 CR, complete response: disappearance of all lesions; PD, disease progression: ≥10% increase in target lesion size and does not meet tumor density criteria of PR density; PR, partial response: ≥10% decrease in target lesion size or ≥15% decrease in tumor density; SD, stable disease: none of the CR, PR, or PD criteria met; RECIST, Response Evaluation Criteria in Solid Tumors
Time Frame: At baseline and every other cycle (± 1 week) until evidence of PD, up to 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Endometrial Cancer | Cervical Cancer
Number analyzed (Participants) | 10 | 7
Participants
  SD ≥ 4 months | 1 | 0
  PD | 9 | 7

3. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) was defined as the time from the date of first infusion of study treatment to the date of progression or death (due to any cause). If progression or death had not occurred at the time of the analysis, PFS was censored on the date of last tumor evaluation.
  PD, disease progression: ≥10% increase in target lesion size and does not meet tumor density criteria of PR density
Time Frame: From the date of first infusion of study treatment to the date of progression or death, up to 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Endometrial Cancer | Cervical Cancer
Number analyzed (Participants) | 10 | 7
months | 1.8 [1.7 to 2.0] | 1.5 [1.5 to 1.8]

4. Secondary Outcome: Progression Free Survival Rate at 4 Months
Description: Progression-free survival rate at 4 months was defined as the percentage of patients who did not progress and were alive at 4 months.
  PD, disease progression: ≥10% increase in target lesion size and does not meet tumor density criteria of PR density
Time Frame: At 4 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Endometrial Cancer | Cervical Cancer
Number analyzed (Participants) | 10 | 7
percentage of participants | 10 [0.0 to 28.6] | 0 [0 to 0]

5. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from the date of first infusion of study treatment to the date of death (due to any cause). Patients with no documented death were censored at the last date they were known to be alive
Time Frame: From the date of first infusion to the date of death, up to 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Endometrial Cancer | Cervical Cancer
Number analyzed (Participants) | 10 | 7
months | 5.5 [4.8 to 11.5] | 5.6 [NA to NA] — Insufficient number of participants with events

6. Secondary Outcome: PM00104 Plasma PK Parameters (Cmax) at First Infusion
Description: Cmax Maximum plasma concentration, directly determined from the experimental data
Time Frame: 0 (Pre-infusion) and 1, 1.5, 3, 7, 24, 48, 168 hours after the end of first infusion (Day 1)
Population: All treated patients
Measure: Mean (Standard Deviation); unit: μg/l
Groups:
- PM00104: Zalypsis (PM00104): Zalypsis (PM00104) (2.5 mg/vial) is provided as a powder for concentrate for solution for infusion
Arm/Group | PM00104
Number analyzed (Participants) | 19
μg/l | 26.47 (11.98)

7. Secondary Outcome: PM00104 Plasma PK Parameters (AUC) at First Infusion
Description: AUC Area under the plasma concentration-time curve from time zero to infinity.
Time Frame: 0 (Pre-infusion) and 1, 1.5, 3, 7, 24, 48, 168 hours after the end of first infusion (Day 1)
Population: All treated patients
Measure: Mean (Standard Deviation); unit: h*μg/l
Arm/Group | PM00104
Number analyzed (Participants) | 19
h*μg/l | 80.88 (37.41)

8. Secondary Outcome: PM00104 Plasma PK Parameters (Cmax) at Second Infusion
Description: Cmax Maximum plasma concentration, directly determined from the experimental data
Time Frame: 0 (Pre-infusion) and 1, 1.5, 3, 7, 24, 48, 168 hours after the end of second infusion (Day 8)
Population: All treated patients with second infusion
Measure: Mean (Standard Deviation); unit: μg/l
Arm/Group | PM00104
Number analyzed (Participants) | 16
μg/l | 35.02 (21.06)

9. Secondary Outcome: PM00104 Plasma PK Parameters (AUC) at Second Infusion
Description: AUC Area under the plasma concentration-time curve from time zero to infinity
Time Frame: 0 (Pre-infusion) and 1, 1.5, 3, 7, 24, 48, 168 hours after the end of second infusion (Day 8)
Population: All treated patients with Second infusion
Measure: Mean (Standard Deviation); unit: h*μg/l
Arm/Group | PM00104
Number analyzed (Participants) | 16
h*μg/l | 86.55 (40.41)

ADVERSE EVENTS:
Time Frame: From first infusion to study termination, up to 2 years
Arm/Group | Endometrial Cancer | Cervical Cancer
All-Cause Mortality (participants affected / at risk) | 9/12 | 5/7
Serious Adverse Events (participants affected / at risk) | 5/12 | 3/7
Other Adverse Events (participants affected / at risk) | 12/12 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endometrial Cancer (N=12) | Cervical Cancer (N=7)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Endocarditis noninfective (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Troponin I increased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Enterobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endometrial Cancer (N=12) | Cervical Cancer (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 4 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (3) | 0 (0)
Vision blurred (Eye disorders) | 2 (3) | 0 (0)
Visual disturbance (Eye disorders) | 2 (3) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 2 (3)
Constipation (Gastrointestinal disorders) | 7 (13) | 5 (13)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (16) | 4 (6)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (6)
Asthenia (General disorders) | 2 (4) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (1)
Chills (General disorders) | 3 (4) | 0 (0)
Fatigue (General disorders) | 7 (15) | 6 (12)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 2 (2)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 5 (8) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (5) | 2 (3)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2010-09-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT00900562/Prot_000.pdf
  • Statistical Analysis Plan (2009-07-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT00900562/SAP_001.pdf